CLINICAL TRIAL: NCT01718067
Title: Efficacy of Vakum Technology in Patients With Chronic Hypersecretion.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Villa Pineta Hospital (Other)
Responsible Party: Principal Investigator, Prof. Clini Enrico, Prof., Villa Pineta Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2793
Record Dates: First submitted 2012-10-22; First posted 2012-10-31 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Bronchitis/Bronchiectasis; Chronic Obstructive Pulmonary Disease
Keywords: Chest physiotherapy; Rehabilitation; Chronic respiratory diseases
MeSH Terms: conditions — Bronchitis, Chronic; Bronchiectasis; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vakum (Experimental): VAKÜM system (Free Aspire, MPR, Legnano-I) added to the conventional manual ELTGOL technique
  Interventions: Device: VAKÜM system; Other: conventional manual ELTGOL technique
- Control (Active Comparator): conventional manual ELTGOL technique
  Interventions: Other: conventional manual ELTGOL technique

INTERVENTIONS:
Device: VAKÜM system — 15 minutes, twice a day.
  Other Names: Free Aspire, MPR, Legnano-I
  Arms: Vakum
Other: conventional manual ELTGOL technique — 20 minutes twice a day

SUMMARY:
Mechanical devices to increase the individual's bronchial hygiene are commonly used to assist patients with chronic retention of secretions. VAKÜM technology has been recently developed with the aim to improve the respiratory condition in hypersecretive patients suffering from chronic respiratory diseases.

The aim of this study is to assess the clinical efficacy of VAKÜM technology in patients with hypersecretion, and chronic respiratory diseases a clinical trial has been designed.

Patients with chronic respiratory diseases, hypersecretion (sputum production >30 mL/die), and reduced cough efficiency (Peak Cough Expiratory Flow > 150 and < 300 L*min-1) referred to standard pulmonary rehabilitation (PR) will be included. Study design is a single-blind multicentre randomized trial with consecutive recruitment. Following a preliminary run-in period, group comparison will be made between Intervention group using VAKÜM system (Free Aspire, MPR, Legnano-I) added to the conventional manual ELTGOL technique, and Control group using manual ELTGOL alone over 10 daily sessions.

Spirometric lung volumes, respiratory muscle strength, arterial blood gases, and quality of life will be recorded in both groups pre-to-post PR. Perceived dyspnea (by VAS scale), sputum volume and characteristics (on a semi-quantitative 3-point scale) and peak expiratory air flows (PEF and PCEF) will be registered on a daily basis over the study period. Primary outcome is the change in perceived dyspnea; in order to ensure 80% power to detect a 5 point (SD 5) group difference change in the primary outcome at the end of the study period as significant at the 0.05 level, at least 42 patients per group are needed. The minimum target sample size will be then fixed at 50 patients per group.

An higher and faster significant reduction of the perceived dyspnea is supposed in the Intervention group. Additional benefits among the secondary outcomes are also hypothesised in the same group.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic respiratory diseases
* hypersecretion condition(sputum production >30 mL/die)
* reduced cough efficiency (Peak Cough Expiratory Flow > 150 and < 300 L*min- 1)
* patients admitted to standard pulmonary rehabilitation

Exclusion Criteria:

* not able to use the device
* concomitant cardiovascular or neoplastic diseases
* utilization of Non Invasive Ventilation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Change in perceived dyspnea | Baseline and 10 days
  Visual Analogic Scale (VAS)

SECONDARY OUTCOMES:
Change in peak expiratory air flows | Baseline and 10 days
  Peak Expiratory Flow (PEF), Peak Cough Expiratory Flow (PCEF)
Change in arterial blood gases exchanges | Baseline and 10 days
  PaO2, PaCO2, SatO2, pH
Change in spirometric lung volumes | Baseline and 10 days
  Static and dynamic lung volumes
Change in respiratory muscle strength | Baseline and 10 days
  Maximal Expiratory Pressure (MEP), Maximal Inspiratory Pressure (MIP)
Change in sputum volume and characteristics | Daily over 10 days
  Volume, Density (D) and Purulence (P) (D and P assessed on a semi-quantitative 3-point scale)
Change in quality of life | Baseline and 10 days
  Quality of life questionnaires (CAT, MRF 28)

CONTACTS AND LOCATIONS:
Overall Officials: Enrico M Clini, MD, Principal Investigator — University of Modena Reggio Emilia
Locations (1):
- Villa Pineta Hospital, Modena, Italy